CLINICAL TRIAL: NCT06117098
Title: Stepping Stones for Successful Evaluation of Mobile App Efficacy for Risk Reduction of Type 2 Diabetes
Brief Title: Mobile App for Risk Reduction of Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 887029
Record Dates: First submitted 2023-05-31; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-03

CONDITIONS: Prediabetic State
Keywords: Prevention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: RCT feasibility study, non-inferiority and superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile application (Experimental): This group will receive individual guidance via the mobile application (12 weeks)
  Interventions: Device: Mobile application
- Group-based lifestyle intervention at the Healthy Lifestyle Centres (Active Comparator): This group will receive a group-based lifestyle intervention program at a Healthy Lifestyle Centre (12 weeks)
  Interventions: Behavioral: Group-based lifestyle intervention
- Group-based lifestyle intervention at a Healthy Lifestyle Centre and recieving a mobile application (Experimental): This group will receive a group-based lifestyle intervention program at a Healthy Lifestyle Centre plus the mobile application (12 weeks)
  Interventions: Behavioral: Group-based lifestyle intervention at a Healthy Lifestyle Centre + mobile application"

INTERVENTIONS:
Device: Mobile application — Individual lifestyle intervention via an mobile application
  Arms: Mobile application
Behavioral: Group-based lifestyle intervention at a Healthy Lifestyle Centre + mobile application" — Group-based lifestyle intervention at a Healthy Lifestyle Centre + mobile application"
  Arms: Group-based lifestyle intervention at a Healthy Lifestyle Centre and recieving a mobile application
Behavioral: Group-based lifestyle intervention — Group-based life style intervention at a Healthy Lifestyle Centre (ususal care)
  Arms: Group-based lifestyle intervention at the Healthy Lifestyle Centres

SUMMARY:
The aim of this feasibility study is to investigate whether a full scale RCT on the efficacy of a mobile app for risk reduction on type 2 diabetes can be conducted in the way it is planned or whether it needs to be modified. This will be investigated through a feasibility study (small scale RCT) on the efficacy of mobile technology on risk reduction of type 2 diabetes.

DETAILED DESCRIPTION:
A small scale RCT will be carried out a the collaborating Healthy Life Centres (HLC). Trained health personnel will deliver the lifestyle programs at these centres, and the content of their programs should be in line with the national guidelines for physical activity and nutrition. The study sample 60 participants with high risk of developing diabetes type 2.

The participants will be randomized into three study arms, 20 participants in each. One group, the intervention group, will receive the mobile app, the second group will receive group-based lifestyle intervention at the HLCs and the third group will receive group based lifestyle intervention at the HLCs and a mobile application. The middle arm will serve as the control arm for both the non-inferiority trial ( mobile application group and HLC lifestyle intervention only) and for the superiority trial (HLC lifestyle intervention plus mobile app and HLC intervention only).

ELIGIBILITY:
Inclusion Criteria:

* smart phone
* prediabetes

Exclusion Criteria:

* not interested in lifestyle change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Six months
  We want to assess the proportion of participants willing and able to take part in the study after referral from general practitioner in two different regions in East Norway. Information will be recorded continuously after telephone contact.
Resources | Nine months
  We will assess the randomization procedure and asses time spent on the first consultation with the participants. Throughout the study period, the supervisor will log all time spent monitoring participants and giving individual feedback through the app.
Management | Nine months
  The use of the app will be registered in terms of actual use and if patients answered tasks within a week, all based on data shown in the administrator interface. Data on adherence to provided tasks and problems experienced with the mobile app will be retrieved from the app-database. We will also assess whether there are any problems with data management involved in the study and assess whether the study personnel had any challenges in conduct of the study.
Satisfaction with the app | Three months
  User satisfaction with the application will be assessed with the System Usability Scale. (SUS), a paper questionnaire at the end of the intervention.The SUS is a technology independent, 10-item questionnaire with a score between 0 and 100 were 0 represents low usability and 100 represent high usability. We will also asses the experienced usefulness of the app after 12 weeks. This will be measured through a questionnaire designed for this study consisting of 16 questions; 13 questions with answers on a Likert scale (0 to 100), 3 multiple-choice questions, and 1 open-ended question.
Change and ceiling and floor effect in outcomes | Three months
  These outcomes will be determined by evaluating whether changes in quality of life and physical activity over a 12-week period could be observed and whether these outcomes disclose ceiling or floor effects. To assess these domains, we will use part of standard questionnaires being used in Healthy Life Centers at the beginning and ending of a 12-week intervention period, being the COOP/WONCA (the Dartmount COOP/World Organization of Family Doctors functional health assessment). This is a questionnaire assessing changes in quality of life.It consists of six questions across six domains with a score of 1 in each domain representing the best possible score while a score of 5 is the worst possible score. Physical activity will be assessed with the validated International Physical Activity Questionnaire (IPAQ) short form. It consists of eight items and encompasses questions regarding time spent walking, in moderate and vigorous intensity physical activity, besides sitting time.

SECONDARY OUTCOMES:
Antropometric measures | Three months
  Weight and waist circumference will be measured at baseline and at the end of the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Blakstad Nilsson, Phd, Principal Investigator — OsloMet
Locations (1):
- OsloMet, Oslo, Norway